CLINICAL TRIAL: NCT00721383
Title: Clinical Trial to Enhance Caregiver Physical Activity
Brief Title: Telephone Resources and Assistance for Caregivers (TRAC)
Acronym: TRAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, Carol J Farran, DNSc, RN, FAAN, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04092307
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Alzheimer's Disease
Keywords: caregiving, Alzheimer's disease, physical activity
MeSH Terms: conditions — Alzheimer Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Physical activity and caregiver skill-building
  Interventions: Behavioral: Enhancing Physical Activity Intervention
- Control (Active Comparator): caregiver skill-building
  Interventions: Behavioral: CSBI

INTERVENTIONS:
Behavioral: Enhancing Physical Activity Intervention — Physical activity and caregiver skill-building
  Other Names: EPAI
  Arms: Treatment
Behavioral: CSBI — Caregiver skill-building
  Arms: Control

SUMMARY:
The purpose of this randomized clinical trial is to test a 12-month multi-component health promotion intervention with home-based family caregivers of persons with Alzheimer's Disease and other related dementias. Specific aims are to: 1) Test the primary hypothesis: The Enhancing Physical Activity treatment intervention will be more effective in increasing caregiver lifestyle physical activity than the Standard Care Intervention; 2) Test secondary hypotheses: The Enhancing Physical Activity treatment intervention will be more effective than the Standard Care Intervention in improving the following caregiver secondary outcomes: mental health, physical health and physical function; and 3) Evaluate the process of implementing a lifestyle physical activity intervention with family caregivers. The Standard Care Intervention focuses on well-established care-related education and support needs. The Enhancing Physical Activity treatment intervention focuses on two areas: increasing lifestyle physical activity and addressing well-established care-related concerns that are likely to interfere with increasing physical activity. A total of 190 middle-age to older community-based primary caregivers of persons with Alzheimer's disease or other related dementias who report some to moderate strain with caregiving activities will be randomly assigned to either the Enhancing Physical Activity or Standard Care Intervention. Data will be collected at baseline, 3, 6, 9, 12 and 18 months and include self-report and direct observational methods. Data will be analyzed by using repeated measures models using the generalized estimating equation approach. Family caregivers are a stressed population who experience changes in their mental and physical health. However, effect sizes have been minimal for interventions designed to only affect caregiver mental health. No study known to us, has tested the added value of physical activity adoption in conjunction with more traditional caregiver support and skill building. Study findings will enable us to evaluate the behavioral , physical, and health-related quality of life effects achieved by the combined intervention; and will add knowledge about the most effective ways of intervening with family caregivers and other chronically stressed middle-age and older adult populations.

ELIGIBILITY:
Inclusion Criteria:

Care recipient:

* Diagnosis of probable AD or related dementia (using NINCDS/ADA criteria)
* Reside in the community
* Receive assistance from a primary caregiver

Caregiver:

* Are a spouse or other close family member of the person with AD/dementia
* Age ≥ 40 years
* English-speaking
* Live with the care recipient (or close as in 5-10 miles)
* Provide ≥ 10 hours of care per week
* Caregiver for at least 6 months
* Are physically inactive, defined as accumulating ≤ 60 minutes of regular PA on a weekly basis for the past 6 months
* Reporting some to moderate levels of strain
* Are cognitively intact
* Have no major debilitating health problems that would prevent intervention participation
* Must have a telephone
* Willing to increase levels of physical activity
* Agree to assignment of treatment condition

Exclusion Criteria:

Care receiver:

* Other dementias such as stroke or Parkinson's
* Terminal illness with life expectancy of less than six months
* Bedfast or confined to a bed or chair at least 22 hours a day for at least 3 of the previous 7 days
* ≥ 3 acute or medical or psychiatric hospitalizations in last year

Caregiver:

* Are involved in another caregiver clinical trial
* Have a terminal illness with life expectancy of less than 6 months
* Receiving active treatment for cancer

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2007-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
self-reported physical activity | 18 months

SECONDARY OUTCOMES:
caregiving burden | 18 months
caregiver positive well-being | 18 months
self-reported physical health | 18 months
physical function | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Farran, PhD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - Rush University Medical Center, Chicago, Illinois